CLINICAL TRIAL: NCT06698861
Title: A Phase 1, Randomized, Open-label Study to Evaluate the Safety, Tolerability, and Pharmacokinetics/Pharmacodynamics of PEG-MetHuG-CSF (P2203) in Healthy Volunteers
Brief Title: A Phase I PK/PD Study of PEG-MetHuG-CSF (P2203) in Healthy Volunteers
Acronym: P2203 phase I
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PharmaEssentia (Industry)
Collaborators: Novotech CRO (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: F23-101
Record Dates: First submitted 2024-10-28; First posted 2024-11-21 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: PK in Healthy Volunteers
Keywords: immunomodulator
MeSH Terms: interventions — pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort 1: PEG-MetHuG-CSF 2 mg (Experimental): To evaluate the safety and tolerability of P2203. In Cohort 1, the first two subjects will be the sentinel subjects treated with staggered dosing. The 1st sentinel subject of Cohort 1 will be dosed at least 96 hours prior to the 2nd sentinel subject. The 2nd sentinel subject will receive P2203 when the Criteria for Dosing Suspension or Termination in a Given Dose Cohort is not met at least during the first 96 hours following administration of P2203 of the 1st sentinel subject. The remaining subject in Cohort 1 will receive P2203 when the Criteria for Dosing Suspension or Termination in a Given Dose Cohort is not met at least during the first 96 hours following administration of P2203 of the 2nd sentinel subject.
  Interventions: Drug: PEG-MetHuG-CSF
- Cohort 2b: Neulasta 6 mg (Active Comparator): In Cohort 2, subjects will be randomized in a 1:1 ratio to receive a single dose of 6 mg P2203 (Cohort 2a, 12 subjects) or a single dose of 6 mg pegfilgrastim (Cohort 2b, 12 subjects).
  Interventions: Drug: Neulasta (Amgen)
- Cohort 2a: PEG-MetHuG-CSF 6 mg (Experimental): In Cohort 2, subjects will be randomized in a 1:1 ratio to receive a single dose of 6 mg P2203 (Cohort 2a, 12 subjects) or a single dose of 6 mg pegfilgrastim (Cohort 2b, 12 subjects).
  Interventions: Drug: PEG-MetHuG-CSF

INTERVENTIONS:
Drug: PEG-MetHuG-CSF — Single dose of PEG-MetHuG-CSF will be given SC injection at 2 mg in Cohort 1 and 6 mg in Cohort 2
  Arms: Cohort 1: PEG-MetHuG-CSF 2 mg; Cohort 2a: PEG-MetHuG-CSF 6 mg
Drug: Neulasta (Amgen) — Single dose of Neulasta will be given SC injection at 6 mg in Cohort 2b.
  Arms: Cohort 2b: Neulasta 6 mg

SUMMARY:
The goal of this study type: PK clinical trial is to evaluate the safety, tolerability, and pharmacokinetics/ pharmacodynamics of PEG-MetHuG-CSF (P2203) in Healthy Volunteers.

Primary objective:

‧ To evaluate the safety and tolerability of P2203

Secondary objectives:

‧ To characterize the pharmacokinetics (PK), pharmacodynamics (PD), and immunogenicity of P2203

Approximately 30 healthy volunteers will be enrolled. Subjects will be screened within 28 days before study dosing. Eligible subjects will be sequentially enrolled into 2 escalating-dose cohorts (Cohort 1 and 2) to receive a single dose of P2203 at a pre-determined specific dose or to re-ceive a single dose of 6 mg pegfilgrastim (Neulasta).

DETAILED DESCRIPTION:
Subjects will be sequentially enrolled into the following inter-subject dose escalation cohorts:

* Cohort 1 (6 subjects): single dose of P2203 at 2 mg
* Cohort 2 (24 subjects): subjects in Cohort 2 will be randomized in a 1:1 ratio to receive a single dose of 6 mg P2203 (Cohort 2a, 12 sub-jects) or a single dose of 6 mg pegfilgrastim (Cohort 2b, 12 subjects).

In Cohort 1, the first two subjects will be the sentinel subjects treated with staggered dosing. The 1st sentinel subject of Cohort 1 will be dosed at least 96 hours prior to the 2nd sentinel subject. The 2nd sentinel subject will receive P2203 when the Criteria for Dosing Suspension or Termination in a Given Dose Cohort (Section 3.5) is not met at least during the first 96 hours following administration of P2203 of the 1st sentinel subject. The remaining subject in Cohort 1 will receive P2203 when the Criteria for Dosing Suspension or Termination in a Given Dose Cohort is not met at least during the first 96 hours following administration of P2203 of the 2nd sentinel subject.

In Cohort 2a, the first three subjects will be the sentinel subjects treated with staggered dosing. The rule and time interval for the stagger dosing in the sentinel subjects in Cohort 2a are the same as those in Cohort 1.

In Cohort 2, subjects will be randomized in a 1:1 ratio to receive a single dose of 6 mg P2203 (Cohort 2a, 12 subjects) or a single dose of 6 mg pegfilgrastim (Cohort 2b, 12 subjects).

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and voluntarily sign an informed consent form (ICF);
2. Age ≥18 and ≤45 years of age at the time of informed consent;
3. Subjects with a body weight ≥ 50 kg and with a body mass index (BMI) of ≥18.5 and <30 kg/m2;
4. Subjects who are non-smokers for at least 24 weeks preceding Screening;
5. Males and females of childbearing potential, as well as all women <2 years after the onset of menopause, must agree to use effective methods of contraception during the entire study period and for 12 weeks after dosing on Day 1; and females must agree to not breastfeed during the study;
6. Subjects who are healthy as determined by pre-study medical his-tory, physical examination, and 12-lead ECG;
7. Subjects whose clinical laboratory test results are within the refer-ence ranges for hematological parameters at Screening and admis-sion (Day -1 or Day 1 pre-dose). All other clinical laboratory test results must be within the reference range or judged not to be clini-cally significant and acceptable to the Investigator.

Exclusion Criteria:

1. Clinically significant illness or surgery within 28 days prior to Dosing;
2. Subjects have previously received G-CSF-related products;
3. Donation of blood or any blood loss > 500 mL in the last 12 weeks prior to Screening;
4. Clinically significant vital sign abnormalities after ≥ 5 minutes supine or sitting rest, defined as any of the following values at Screening or admission (Day -1):

   * systolic blood pressure <90 or ≥ 140 mmHg; or
   * diastolic blood pressure <50 or ≥ 90 mmHg; or
   * pulse rate <50 or >100 beats per minutes.
5. Subjects who have any clinically important abnormalities in the 12-lead ECG at Screening as considered by the Investigators that may pose a risk to subjects or interfere with the interpretation of QTc interval changes;
6. Subjects who have a prolonged QTcF >450 ms at Screening or family history of long QT syndrome;
7. Subjects with history of drug or alcohol abuse; or those with positive result in the drug or ethanol examination at Screening or admission (Day -1);
8. Subjects who are positive for hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab), or human immunodeficiency virus (HIV) antibody at Screening;
9. Subjects with latex hypersensitivity or those have a history of severe allergy and/or severe drug reaction (e.g., anaphylaxis, other drug reaction requiring hospitalization, OR any other drug hypersensitivity); or those have known allergic reactions to any component of the treatments in this study;
10. Immunization with a live attenuated vaccine during a 28-day period prior to dosing, immunization with an inactivated or mRNA vaccine during a 14-day period prior to dosing, or planned immunization of any kind of vaccine during the course of the study;
11. Subjects with syphilis or those have a clinically significant history or evidence of any active or suspected bacterial, viral, fungal or parasitic infection, or unexplained cause of clinically significant inflammatory, within the 28 days prior to Dosing, e.g., common cold, viral syndrome, flu-like symptoms, etc;
12. Subjects who have acute gastrointestinal symptoms at Screening or admission (Day -1) (e.g., nausea, vomiting, diarrhea, and heartburn);
13. Take any prescription drugs within 14 days or nonprescription drugs (except routine vitamins at the recommended daily dose) within 7 days prior to Dosing were not allowed unless specified in the protocol or agreed as not clinically relevant by the Principal Investigator;
14. History of body organ transplant and are taking immunosuppressants at Screening; subject with history of bone marrow/hematopoietic stem cell transplantation, regardless of whether s/he is taking immunosuppressants at Screening, will be excluded;
15. Subjects who have received other investigational product within the last 12 weeks or within 5 times the half-life prior to Screening, whichever is longer;
16. Subjects who have received drugs containing lithium, systemic immunosuppressants, e.g., corticosteroid, or herbal remedies within 28 days prior to screening;
17. Subjects who have consumed grapefruit, grapefruit juice or other products containing grapefruit within 7 days prior to Dosing;
18. History of any malignant disease, including solid tumor and hematologic malignancies;
19. Pregnant subjects;
20. Subjects who are unlikely to co-operate with the requirements of the study;
21. Any reason which, in the opinion of the investigator, would prevent the subject from participating in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-08-19 (Actual); Primary Completion 2025-02-06 (Actual); Study Completion 2025-02-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of P2203 injection. | from day 1 to day 36
  The safety and tolerability of P2203 injection are evaluated by the occurrence of the adverse events, serious adverse events, and the abnormal clinical laboratory data, ECG changes, physical examination findings, and lab examinations.
To determine the maximum tolerated dose of P2203 | from Day 1 to Day 29
  The maximum tolerated dose is defined as the highest tolerated dose level without the occurrence of predetermined unacceptable safety scenario during the 28-day safety monitoring period. Unacceptable safety scenario includes:
  * ≥ 1 of 6 subjects in Cohort 1 or ≥ 1 of 12 subjects in Cohort 2a experiences SAE(s) which is at least possibly related to P2203;
  * ≥ 2 of 6 subjects in Cohort 1 or ≥ 2 of 12 subjects in Cohort 2a have severe (Grade 3 or higher as per CTCAE) non-serious adverse events which is at least possibly related to P2203;
  * ≥ 2 of 6 subjects in Cohort 1 or ≥ 2 of 12 subjects in Cohort 2a have a drug related QTc pro-longation defined as QTcF > 500 ms, or an increase of QTcF > 60 ms above baseline on the 12-lead electrocardiogram (ECG), confirmed (persistent for > 5 minutes) on repeated 12-lead ECGs;
  * The occurrence of significant safety events that may pose a risk to subjects as judged by the SRC review; any adverse event(s) leading to subject withdrawal must be judged b

CONTACTS AND LOCATIONS:
Locations (1):
- Mackay Memorial Hospital, Taipei, Taiwan, Taipei, Taiwan, Taiwan